CLINICAL TRIAL: NCT01435408
Title: A Randomised Comparison of the Clinical Outcome After Postconditioning or Deferred Stent Implantation Versus Conventional Treatment
Brief Title: DANish Study of Optimal Acute Treatment of Patients With ST-elevation Myocardial Infarction
Acronym: DANAMI-3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Engstrom, MD, DMSci, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DANAMI-3
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: ST Segment Elevation Myocardial Infarction
Keywords: STEMI; Ischemic postconditioning; Deferred stenting; Primary PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ischemic Postconditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional treatment. (Active Comparator): Conventional primary PCI in STEMI.
  Interventions: Other: Conventional primary PCI
- IPost (Experimental): Ischemic postconditioning in STEMI.
  Interventions: Other: Ischemic postconditioning.
- Deferred primary PCI. (Experimental): Deferred strategy in STEMI.
  Interventions: Other: Deferred stenting in primary PCI.

INTERVENTIONS:
Other: Conventional primary PCI — Conventional primary PCI in STEMI with implantation of DES.
  Other Names: pPCI
  Arms: Conventional treatment.
Other: Ischemic postconditioning. — Primary PCI in STEMI with implantation of DES. Following re-opening of the culprit artery mechanical postconditioning with 4 cycles of 30/30 sec. reperfusion/re-occlusion i performed.
  Other Names: Ischemic postconditioning; Mechanical postconditioning
  Arms: IPost
Other: Deferred stenting in primary PCI. — In STEMI re-opening of the artery with guidewire/thrombectomy/small size balloon inflation DES stenting is postponed for 48 hours.
  Other Names: Deferred stenting
  Arms: Deferred primary PCI.

SUMMARY:
This study focuses on Cardioprotective strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Acute onset of chest pain of < 12 hours' duration.
* ST-segment elevation ≥ 0.1 mV in ≥ 2 contiguous leads, signs of a true posterior infarction or documented newly developed left bundle branch block.

Culprit lesion in a major native vessel.

Exclusion Criteria:

* Pregnancy.
* Known intolerance of ASA, clopidogrel, heparin or contrast.
* Inability to understand information or to provide informed consent.
* Haemorrhagic diathesis or known coagulopathy.
* Stent thrombosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2011-04; Primary Completion 2016-02 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
All cause mortality, heart failure (postconditioning) | 2 years

SECONDARY OUTCOMES:
Infarct size in relation to area at risk as determined by MRI after 3 month | 3 month
  Infarct size Salvage index
All cause mortality, myocardial infarction, repeat revascularisation and occurrence of definite stent thrombosis according to ARC definition within 1 year (deferred stent strategy) | 1 year

OTHER OUTCOMES:
TIMI flow | postprocedure
ST-segment resolution | 90 min postprocedure
Wall motion index (echo) | 1 year
LVEF (MRI) | 90 days
Infarct size (MRI) | 90 days
Microvascular obstruction (MVO) | within 48 hours
Quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lars Koeber, Prof., DMSci, Principal Investigator — The Heart Center, Rigshospitalet, University of Copenhagen; Thomas Engstrom, MD, DMSci, Principal Investigator — The Heart Center, Rigshospitalet, University of Copenhagen; Henning Kelbaek, MD, DMSci, Principal Investigator — The Heart Center, Rigshospitalet, University of Copenhagen
Locations (5):
- Denmark (5):
  - Department of Cardiology, Aalborg University Hospital, Aalborg
  - Department of Cardiology, Skejby University Hospital, Aarhus
  - The Heart Center, Rigshospitalet, University of Copenhagen, Copenhagen
  - Department of Cardiology, Gentofte University Hospital, Hellerup
  - Department of Cardiology, Odense University Hospital, Odense

REFERENCES:
- [Derived] Elezi B, Marquard JM, Kelbaek H, Nepper-Christensen L, Ahtarovski K, Kyhl K, Goransson C, Islam U, Kober L, Hofsten D, Pedersen F, Vejlstrup NG, Holmvang L, Engstrom T, Lonborg JT. Ten-year prognostic impact of cardiac magnetic resonance endpoints in patients with ST-segment elevation myocardial infarction. Eur Heart J Cardiovasc Imaging. 2026 Jan 6:jeag001. doi: 10.1093/ehjci/jeag001. Online ahead of print. PMID 41493904
- [Derived] Marquard JM, Engstrom T, Kelbaek H, Beske RP, Islam U, Hofsten DE, Holmvang L, Pedersen F, Terkelsen CJ, Hoj Christiansen E, Tilsted HH, Glinge C, Jabbari R, Eftekhari A, Raungaard B, Clemmensen P, Botker HE, Jensen LO, Kober L, Lonborg JT. 10-Year Outcomes of Deferred or Conventional Stent Implantation in Patients With STEMI (DANAMI-3-DEFER). Circ Cardiovasc Interv. 2025 Jun;18(6):e015369. doi: 10.1161/CIRCINTERVENTIONS.125.015369. Epub 2025 May 20. PMID 40391569
- [Derived] Mazhar J, Ekstrom K, Kozor R, Grieve SM, Nepper-Christensen L, Ahtarovski KA, Kelbaek H, Hofsten DE, Kober L, Vejlstrup N, Vernon ST, Engstrom T, Lonborg J, Figtree GA. Cardiovascular magnetic resonance characteristics and clinical outcomes of patients with ST-elevation myocardial infarction and no standard modifiable risk factors-A DANAMI-3 substudy. Front Cardiovasc Med. 2022 Aug 3;9:945815. doi: 10.3389/fcvm.2022.945815. eCollection 2022. PMID 35990971
- [Derived] Ekstrom K, Nielsen JVW, Nepper-Christensen L, Ahtarovski KA, Kyhl K, Goransson C, Bertelsen L, Ghotbi AA, Kelbaek H, Hofsten DE, Kober L, Schoos MM, Vejlstrup N, Lonborg J, Engstrom T. Ischemia From Nonculprit Stenoses Is Not Associated With Reduced Culprit Infarct Size in Patients with ST-Segment-Elevation Myocardial Infarction. Circ Cardiovasc Imaging. 2021 May;14(5):e012290. doi: 10.1161/CIRCIMAGING.120.012290. Epub 2021 May 5. PMID 33951923
- [Derived] Nepper-Christensen L, Hofsten DE, Helqvist S, Lassen JF, Tilsted HH, Holmvang L, Pedersen F, Joshi F, Sorensen R, Bang L, Botker HE, Terkelsen CJ, Maeng M, Jensen LO, Aaroe J, Kelbaek H, Kober L, Engstrom T, Lonborg J. Interaction of ischaemic postconditioning and thrombectomy in patients with ST-elevation myocardial infarction. Heart. 2020 Jan;106(1):24-32. doi: 10.1136/heartjnl-2019-314952. Epub 2019 Jul 17. PMID 31315939
- [Derived] Ekstrom K, Nepper-Christensen L, Ahtarovski KA, Kyhl K, Goransson C, Bertelsen L, Ghotbi AA, Kelbaek H, Helqvist S, Hofsten DE, Kober L, Schoos MM, Vejlstrup N, Lonborg J, Engstrom T. Impact of Multiple Myocardial Scars Detected by CMR in Patients Following STEMI. JACC Cardiovasc Imaging. 2019 Nov;12(11 Pt 1):2168-2178. doi: 10.1016/j.jcmg.2019.01.032. Epub 2019 Apr 17. PMID 31005537
- [Derived] Nepper-Christensen L, Lonborg J, Hofsten DE, Ahtarovski KA, Bang LE, Helqvist S, Kyhl K, Kober L, Kelbaek H, Vejlstrup N, Holmvang L, Engstrom T. Benefit From Reperfusion With Primary Percutaneous Coronary Intervention Beyond 12 Hours of Symptom Duration in Patients With ST-Segment-Elevation Myocardial Infarction. Circ Cardiovasc Interv. 2018 Sep;11(9):e006842. doi: 10.1161/CIRCINTERVENTIONS.118.006842. PMID 30354595
- [Derived] Falkentoft AC, Rorth R, Iversen K, Hofsten DE, Kelbaek H, Holmvang L, Frydland M, Schoos MM, Helqvist S, Axelsson A, Clemmensen P, Jorgensen E, Saunamaki K, Tilsted HH, Pedersen F, Torp-Pedersen C, Kofoed KF, Goetze JP, Engstrom T, Kober L. MR-proADM as a Prognostic Marker in Patients With ST-Segment-Elevation Myocardial Infarction-DANAMI-3 (a Danish Study of Optimal Acute Treatment of Patients With STEMI) Substudy. J Am Heart Assoc. 2018 May 18;7(11):e008123. doi: 10.1161/JAHA.117.008123. PMID 29776961
- [Derived] Lonborg J, Engstrom T, Ahtarovski KA, Nepper-Christensen L, Helqvist S, Vejlstrup N, Kyhl K, Schoos MM, Ghotbi A, Goransson C, Bertelsen L, Holmvang L, Pedersen F, Jorgensen E, Saunamaki K, Clemmensen P, De Backer O, Klovgaard L, Hofsten DE, Kober L, Kelbaek H; DANAMI-3 Investigators. Myocardial Damage in Patients With Deferred Stenting After STEMI: A DANAMI-3-DEFER Substudy. J Am Coll Cardiol. 2017 Jun 13;69(23):2794-2804. doi: 10.1016/j.jacc.2017.03.601. PMID 28595694
- [Derived] Topal DG, Lonborg J, Ahtarovski KA, Nepper-Christensen L, Helqvist S, Holmvang L, Pedersen F, Clemmensen P, Saunamaki K, Jorgensen E, Kyhl K, Ghotbi A, Schoos MM, Goransson C, Bertelsen L, Hofsten D, Kober L, Kelbaek H, Vejlstrup N, Engstrom T. Association Between Early Q Waves and Reperfusion Success in Patients With ST-Segment-Elevation Myocardial Infarction Treated With Primary Percutaneous Coronary Intervention: A Cardiac Magnetic Resonance Imaging Study. Circ Cardiovasc Interv. 2017 Mar;10(3):e004467. doi: 10.1161/CIRCINTERVENTIONS.116.004467. PMID 28264870
- [Derived] Engstrom T, Kelbaek H, Helqvist S, Hofsten DE, Klovgaard L, Clemmensen P, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, Ravkilde J, Tilsted HH, Villadsen A, Aaroe J, Jensen SE, Raungaard B, Botker HE, Terkelsen CJ, Maeng M, Kaltoft A, Krusell LR, Jensen LO, Veien KT, Kofoed KF, Torp-Pedersen C, Kyhl K, Nepper-Christensen L, Treiman M, Vejlstrup N, Ahtarovski K, Lonborg J, Kober L; Third Danish Study of Optimal Acute Treatment of Patients With ST Elevation Myocardial Infarction-Ischemic Postconditioning (DANAMI-3-iPOST) Investigators. Effect of Ischemic Postconditioning During Primary Percutaneous Coronary Intervention for Patients With ST-Segment Elevation Myocardial Infarction: A Randomized Clinical Trial. JAMA Cardiol. 2017 May 1;2(5):490-497. doi: 10.1001/jamacardio.2017.0022. PMID 28249094
- [Derived] Nepper-Christensen L, Lonborg J, Ahtarovski KA, Hofsten DE, Kyhl K, Ghotbi AA, Schoos MM, Goransson C, Bertelsen L, Kober L, Helqvist S, Pedersen F, Saunamaki K, Jorgensen E, Kelbaek H, Holmvang L, Vejlstrup N, Engstrom T. Left Ventricular Hypertrophy Is Associated With Increased Infarct Size and Decreased Myocardial Salvage in Patients With ST-Segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention. J Am Heart Assoc. 2017 Jan 9;6(1):e004823. doi: 10.1161/JAHA.116.004823. PMID 28069574
- [Derived] Kelbaek H, Hofsten DE, Kober L, Helqvist S, Klovgaard L, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, De Backer O, Bang LE, Kofoed KF, Lonborg J, Ahtarovski K, Vejlstrup N, Botker HE, Terkelsen CJ, Christiansen EH, Ravkilde J, Tilsted HH, Villadsen AB, Aaroe J, Jensen SE, Raungaard B, Jensen LO, Clemmensen P, Grande P, Madsen JK, Torp-Pedersen C, Engstrom T. Deferred versus conventional stent implantation in patients with ST-segment elevation myocardial infarction (DANAMI 3-DEFER): an open-label, randomised controlled trial. Lancet. 2016 May 28;387(10034):2199-206. doi: 10.1016/S0140-6736(16)30072-1. Epub 2016 Apr 3. PMID 27053444
- [Derived] Hofsten DE, Kelbaek H, Helqvist S, Klovgaard L, Holmvang L, Clemmensen P, Torp-Pedersen C, Tilsted HH, Botker HE, Jensen LO, Kober L, Engstrom T; DANAMI 3 Investigators. The Third DANish Study of Optimal Acute Treatment of Patients with ST-segment Elevation Myocardial Infarction: Ischemic postconditioning or deferred stent implantation versus conventional primary angioplasty and complete revascularization versus treatment of culprit lesion only: Rationale and design of the DANAMI 3 trial program. Am Heart J. 2015 May;169(5):613-21. doi: 10.1016/j.ahj.2015.02.004. Epub 2015 Feb 14. PMID 25965708